CLINICAL TRIAL: NCT05489107
Title: New Option for the Treatment of Radiation-induced Proctitis Study
Brief Title: New Local Treatment of Radiation-induced Proctitis
Acronym: NOTRIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Barmherzige Brüder Vienna (Other)
Responsible Party: Principal Investigator, ILIYAN ILIEV, Principal Investigator, General Surgeon, Barmherzige Brüder Vienna
Other Study IDs: 202207-01
Record Dates: First submitted 2022-08-02; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Radiation Proctitis
Keywords: radiation; proctitis; hyaluronic acid; chondroitin sulfate; poloxamer 407; local treatment; rectoscopy
MeSH Terms: conditions — Proctitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ziverel — Within a first flexible rectoscopy (Day 1) the product will be applied transanally. Then the patients will apply it as enemas twice daily for 7 days. On day 8 (after treatment completion), and on day 31 (after 23 days of no treatment) follow-up flexible rectoscopies will be performed.

SUMMARY:
A prospective single-center observational study to evaluate the effectiveness of a local treatment with a mixture of hyaluronic acid, chondroitin sulfate and poloxamer 407 in patients with radiation-induced proctitis.

ELIGIBILITY:
Inclusion Criteria:

* proven symptomatic acute or chronic radiation-induced proctitis;
* current or prior radiation therapy in the pelvic area;
* patients with complications connected to the radiation therapy.

Exclusion Criteria:

* lack of informed consent;
* non-adherence to study protocol;
* pregnancy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 18 and 99 years of age with radiation proctitis under/after prior radiation therapy beacuse of oncological conditions in the pelvic area.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Petechiae in the most affected areas of the rectal mucosa. | 1 month
  Assessment of the effects of the mixture on the number of petechiae in the rectum. Within the first flexible rectoscopy (Day 1) the most affected areas of the rectal mucosa (on the anterior and posterior wall) will be determined. A 27 mm CAPTIVATOR hexagonal polypectomy snare (Boston Scientific) will be introduced through the endoscope, and will be fully opened. The fully open polypectomy snare (9,2 cm2) will be applied over the most affected areas on the anterior and posterior rectal wall, and the number of the petechiae within these areas will be documented. The flexible rectoscopy will be repeated on day 8 after patients have already received enemas with the examined substance twice daily for one week, and the number of the petechiae will be documented as above mentioned. After a period of 23 days with no treatment, a follow-up flexible rectoscopy will be performed on day 31, and the petechiae of the rectal mucosa will be once more assessed.

SECONDARY OUTCOMES:
Assessment of patients' quality of life using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Proctitis Module with 20 Questions (EORTC QLQ-PRT20) | 6 months
  The effects of the mixture on subjects' quality of life will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Proctitis Module with 20 Questions Score (EORTC QLQ-PRT20). The questionnaire consists of 18 quantitative, 2 qualitative (one of them being optional), and 1 semi-quantitative questions . Using the quantitative questions, a score can be defined. Its minimum value is 18 (meaning patients have no symptoms), and its maximum value is 72 (meaning greatest extent of lifestyle limitations because of radiation proctitis). The semi-quantitative question provides information about the highest number of defecations per 24 hours and is not included in the score. The qualitative questions determine the use of medicines, and patients' will to receive any assistance concerning their symptoms.
  The score will be documented on day 1, 8, 31 and 6 months after treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Dauser, Assoc. Prof., Study Chair — Krankenhaus der Barmherzige Brüder Wien
Locations (1):
- Krankenhaus der Barmherzigen Brüder, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No